CLINICAL TRIAL: NCT07021885
Title: Nutrition Literacy and Associated Outcomes in Head and Neck Cancer Survivor-caregiver Dyads
Brief Title: NLit and Outcomes in HNC Survivor-Caregiver Dyads
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: COE Pilot 2023
Record Dates: First submitted 2025-05-29; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Caregiver Burden; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Head and Neck Neoplasms; Caregiver Burden; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational (cross-sectional) study is to better understand nutrition literacy in survivor-caregiver dyads and its impact on nutrition related outcomes and quality of life. We're interested in finding out how much they know about nutrition and how this might relate to their overall health, body composition, functional status, and overall well-being. We will target post-treatment head and neck cancer survivors and a paired informal caregiver.

The main questions we aim to answer are:

* How does the nutrition literacy of both the survivor and caregiver relate to their sociodemographic, behavioral, and clinical characteristics?
* How dyadic nutrition literacy influence individual nutrition outcomes like skin carotenoid levels, body composition, and functional status?
* Does the shared nutrition knowledge (nutrition literacy) of both the survivor and caregiver impact their quality of life together?

Participants will:

Answer questions about their knowledge of nutrition. Have their nutritional health status checked. Use a non-invasive device to measure skin carotenoid content to validate self-reports of fruit and vegetable intake.

Have a simple and painless test to measure their body composition - like how much muscle and fat they have.

Do some physical tests like grip strength and walking to measure their physical ability.

Answer questions about their general well-being and lifestyle, like exercise and diet.

(For the survivor) Share details about their cancer, its treatment, and their overall well-being.

(For the caregiver) Answer questions about their role in taking care of the survivor, and their involvement in care routine such as food shopping and cooking.

ELIGIBILITY:
Inclusion Criteria:

* Survivors and their caregivers will be eligible to participate if the survivor 1) has a history of oral cavity, pharyngeal, or laryngeal cancer, 2) is between 6 months - 4 years post-primary oncology treatment, 3) has no evidence of disease, 4) has an informal caregiver living in or out of the home who has a shared or primary role in food procurement and/or preparation, 5) no current use of feeding tube as the primary source of nutrition and can consume food orally, 6) age 18+, 7) English-speaking. Survivors and their caregivers will not be eligible to participate if either has 1) dementia or organic brain syndrome; 2) severe emotional distress; 3) active schizophrenia, 4) another diagnosis of cancer in the past five years (not including skin or cervical cancer in situ).

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: post-treatment head and neck cancer survivors and a paired informal caregiver
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-08-16 (Estimated); Study Completion 2026-05-16 (Estimated)

PRIMARY OUTCOMES:
Nutrition Literacy | at a single time point between 6 months and 5 years post-treatment
  Measured by the self-administered Nutrition Literacy Assessment Instrument (NLit).
Nutrition Status | at a single time point between 6 months and 5 years post-treatment
  Measured by the Mini Nutrition Assessment (MNA)
Skin Carotenoid | at a single time point between 6 months and 5 years post-treatment
  Using the Veggie Meter®
Body composition | at a single time point between 6 months and 5 years post-treatment
  Measured by BIA - InBody© 270, USA
Functional status | at a single time point between 6 months and 5 years post-treatment
  Handgrip strength will be measured and recorded 3 times using the Jamar hand dynamometer on the dominant hand; Functional performance status will also be assessed using a short physical performance battery consisting of three functional tests assessing performance.
Sociodemographics. | at a single time point between 6 months and 5 years post-treatment
  Age, biological sex, race, ethnicity, years of education, annual household income, employment status, pack-years smoking, alcohol consumption (current, former, never) will be self-reported.
Fruit & Vegetable Intake | at a single time point between 6 months and 5 years post-treatment
  Using the Eating at America's Table Study's (EATS) All-Day screener designed, and validated by the National Cancer Institute
Exercise | at a single time point between 6 months and 5 years post-treatment
  Assessed using a modified Godin Leisure-Time Exercise Questionnaire
Food Security | At a single time point between 6 months and 5 years post-treatment
  Self-reported food security will be assessed using the USDA's U.S. Household Food Security Survey Module: Six-Item Short Form
Caregiving characteristics | between 6 months and 5 years post-treatment
  Caregiver only: Caregivers will be asked to self-report their residence (in or out of survivor's home), years spent caregiving, hours per week spent caregiving, relationship to survivor, and role in food procurement and preparation
Quality of life | between 6 months and 5 years post-treatment
  Caregiver: Overall quality of life will be assessed using the Caregiver FACT-General, which is structured and scored similarly to the FACT-HN but adapted for use in cancer caregivers. Cancer survivor: Overall quality of life will be assess using the Functional Assessment of Cancer Therapy - Head and Neck (FACT-HN) quality of life questionnaire.
Clinical characteristics | between 6 months and 5 years post-treatment
  Tumor site, cancer stage, treatment modality, and HPV-status of the tumor will be collected through EMR review

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States